CLINICAL TRIAL: NCT03428880
Title: Ultrasound Guided Quadratus Lumborum Type III Block Versus Intrathecal Morphine for Analgesia After Cesarean Delivery
Brief Title: Ultrasound Guided QLB III Versus Intrathecal Morphine for Analgesia After Cesarean Section
Acronym: QLB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Ben marzouk Sofiene, MD, assistant professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: fel-bich
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Block
Keywords: quadratus lumborum block; cesarean section; spinal morphine; ultrasound guidance
MeSH Terms: conditions — Bites and Stings | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- spinal morphine (Active Comparator): intrathecal morphine with 10 mg bupivacaine, 5 gamma sufenta and 100 gamma morphine. Intervention: In the end of surgery a QLB block is done with 20 ml of normal saline per side.
  Interventions: Drug: Morphine
- quadratus lumborum block (Active Comparator): intrathecal anesthesia with10 mg bupivacaine, 5 gamma sufena and 1 ml normal saline.
  Procedure : a quadratus lumborum block is done with 20 ml of bupivacaine 0,125% per side.
  Interventions: Drug: Quadratus lumborum block

INTERVENTIONS:
Drug: Morphine — spinal morphine is done before cesarean section
  Other Names: spinal morphine
  Arms: spinal morphine
Drug: Quadratus lumborum block — a US Block QLB is done after surgery
  Other Names: QLB
  Arms: quadratus lumborum block

SUMMARY:
Subarachnoid morphine (SAM) is the gold standard for treating postoperative pain after cesarean delivery (CD) but it has undesirable side effects, that's why the aim of our study is to identify whether ultrasound-guided Quadratus lumborum block type 3, a new regional anesthetic technique that blocks the abdominal wall neural afferents, can provide at the same time better postoperative analgesia after CD with less side effects

DETAILED DESCRIPTION:
In this prospective double blinded randomized study,120 parturients undergoing cesarian delivery via a Pfannenstiel incision and who agreed to spinal anesthesia were randomly scheduled to receive either a SAM (group SAM, n=60) or a Quadratus lumborum block type 3 (group QLB, n=60).Spinal anesthesia was initiated with hyperbaric Bupivacaïne 0.5% 10 mg, 0,005 mg SUFENTANIL MEDIS and 0.1 mg morphine in the SAM group and with Bupivacaïne 0.5% 10 mg, 0,005 mg SUFENTANIL MEDIS and 1 ml normal saline in group QLB.

After surgery, bilateral QLB block type 3 was performed with the patient in lateral position using bupivacaine 0.25% , 20 mL on each side in group QLB and 20 ml normal saline in group SAM.

Postoperative analgesia for the first 24 hours consisted of a patient controlled analgesia with IV morphine only. If necessary breakthrough pain was treated by 01 g paracetamol intravenously by the same doctor in charge of taking the values of the visual analogue scale.

Patients were assessed postoperatively in the postanesthesia care unit (time 0 hours) and at 2, 4, 6, 12 and 24 hours.

Visual analogue scale (VAS) for pain at rest and during the palpation of the uterine globe was noted.

The primary outcome measure was the total dose of morphine over 24 hours delivered by a patient-controlled analgesia system at predetermined intervals.

Secondary outcomes were visual analogue scale (VAS) for pain at rest and on the palpation of the uterine globe ,heart rate, blood pressure, itching, nausea, pruritus, vomiting and sedation.

ELIGIBILITY:
Inclusion Criteria:

* ASA I/II.
* Normal singleton pregnancy with a gestation of at least 37 weeks.

Exclusion Criteria:

* Heart disease
* Coagulopathy
* pre-eclampsia
* BMI> 40
* Patient refusal to undergo the Quadratus lumborum block.
* Allergy to local anesthetics

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption over 24 hours postoperatively | Arrival to post anesthesia care unit until 24 hours posteratively
  Total IV morphine used when started postoperatively using a PCA with morphine in the post anesthesia care unit until 2' hours posteratively.

SECONDARY OUTCOMES:
Time to first analgesic demand using PCA pump with morphine | Arrival to post anesthesia care unit until 24 hours posteratively
  recording the exact time to first analgesic demand by using the PCA with Morphine
Visual analog scale (VAS) pain scores at rest and during the palpation of the uterine globe | Arrival to post anesthesia care unit until 24 hours posteratively
  At predetermined intervalls, visual analog scale (VAS) pain scores at rest and at the palpation of the uterine globe were noted.
Time to first deambulaton after surgery | Arrival to post anesthesia care unit until 24 hours posteratively
  After surgery, time when the patient was able to move from bed was noted.

CONTACTS AND LOCATIONS:
Overall Officials: Hayene Maghrebi, Professor, Study Chair — tunis maternity center
Locations (2):
- Tunisia (2):
  - Tunis maternity and neonatology center, minisetry of public health, Tunis
  - Tunis maternity and neonatology center,, Tunis

IPD SHARING:
Plan to Share IPD: Undecided